CLINICAL TRIAL: NCT05738213
Title: Hormonal Effects of Puberty-Related Alterations on Pain in Adolescents With Migraine
Brief Title: Puberty, Sex Hormones and Pain Sensitivity in Adolescents With Migraine
Acronym: IHS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: International Headache Society (Unknown)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202208057; Seed Pediatric Research Grant (Other Grant/Funding Number: International Headache Society)
Record Dates: First submitted 2022-12-06; First posted 2023-02-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: pain; puberty; sex hormones
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — carboxypeptidase M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine (Active Comparator): Adolescents with a migraine diagnosis
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Pressure pain thresholds (PPT); Behavioral: Conditioned pain modulation (CPM) response; Behavioral: PedMIDAS (Pediatric Migraine Disability Assessment); Diagnostic Test: Hormonal assessment; Other: Pubertal status
- Healthy control (Placebo Comparator): Adolescents without a migraine diagnosis
  Interventions: Device: Thermal stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Pressure pain thresholds (PPT); Behavioral: Conditioned pain modulation (CPM) response; Diagnostic Test: Hormonal assessment; Other: Pubertal status

INTERVENTIONS:
Device: Thermal stimuli — The Thermal Sensory Analyzer (TSA-II or PATHWAY platform - Medoc, Ramat Yishai, Israel) will be used to safely deliver heat and cold stimuli. These devices can deliver relatively complex stimuli via computer control. All targeted stimulus temperatures will be less than 50°C, and participants will be free to remove their arm or leg at any time from the thermode. Noxious cold stimuli will also be delivered with a plastic water container or a water bath (FISHER, USA). Participants will be free to pull out of the water bath at any time.
  Other Names: Thermal Sensory Analyzer (TSA-II or PATHWAY platform - Medoc, Ramat Yishai, Israel)
Device: Pressure stimuli — Pressure stimuli will be applied by using a handheld algometer (Wagner Instruments) or the Pressure Algometer (Medoc, Ramat Yishai, Israel). These devices have a round probe that allows quantifying the amount of pressure that is being applied. The Pressure Algometer allows a real-time visual feedback to control and monitor applied pressure rates. Pressure will be applied to the lower leg, volar forearm, or trapezius.
  Other Names: handheld algometer (Wagner Instruments); the Pressure Algometer (Medoc, Ramat Yishai, Israel)
Behavioral: Pain ratings — Pain intensity and pain unpleasantness ratings will be assessed.
  Other Names: Numerical rating scale (ranging from 0- no pain/unpleasantness to- 100 the most intense/unpleasantness pain imaginable); mechanical and computerized visual analog scales (VAS which ranges between ''no pain sensation'' and ''most intense pain imaginable'')
Behavioral: Pressure pain thresholds (PPT) — Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements.
Behavioral: Conditioned pain modulation (CPM) response — The CPM paradigm assesses endogenous inhibitory pain modulation efficiency. CPM testing includes the application of a "test" stimulus without conditioning (control run, pressure pain thresholds) and a subsequent application of the same test stimulus together with a conditioning stimulus (conditioning run, a 60 second of foot immersion in cold water). The CPM response is the difference in the pressure pain thresholds between the control and the conditioning runs.
Behavioral: PedMIDAS (Pediatric Migraine Disability Assessment) — Adolescents with migraine will complete questions regarding their headache frequency. Migraine disability will be assessed using PedMIDAS (Pediatric Migraine Disability Assessment). This self-reported questionnaire assesses the number of days that headaches affect participant's daily activities. This is a widely used, reliable and validated tool to assess migraine disability.
  Arms: Migraine
Diagnostic Test: Hormonal assessment — Blood samples (approximetly 2 tablespoons) will be collected for analyses of sex hormone levels (e.g., testosterone, estradiol, progesterone).
Other: Pubertal status — Pubertal status will be assessed using the self-reported Physical Developmental Scale-Wave 3 survey, which allows for differentiation between pre-, early-, late-, and post-pubertal status. Early puberty is defined as a score of 3 and no menarche, mid-puberty is defined as 4 and no menarche, late pubertal is defined as a score of 7 points or less and with menarche, and post pubertal is defined as a score of 8 and menarche. For boys, pubertal maturation status will be determined by the Physical Development Scale using the body hair growth voice change and facial hair questions. Early puberty is defined as a score of 4-5, mid-puberty is defined as a score of 6-8, late pubertal is defined as a score of 9-11 points, and post pubertal is defined as a score of 12.

SUMMARY:
The purpose of this research study is to investigate the relationships between sex hormone levels and experimental pain sensitivity and migraine severity will be examined.

DETAILED DESCRIPTION:
This study will investigate how puberty and variability in sex hormone levels impact pain sensitivity and migraine symptoms.

Hypothesis 1- A significant reduction in pain sensitivity from early to late pubertal status will be found only for adolescents without but not with migraine during pubertal maturation.

Hypothesis 2- Experimental pain sensitivity will be negatively correlated with testosterone levels in adolescents in both groups (with and without migraine).

Exploratory Hypothesis 1- In adolescents with migraine, higher migraine severity (headache frequency and migraine disability) will be associated with lower testosterone levels.

Exploratory hypothesis 2- Adolescents with migraine will have lower testosterone levels than those without.

ELIGIBILITY:
Inclusion criteria

1. Age between 11-15
2. Males and females
3. English speakers
4. Migraine group: diagnosed with migraine
5. Control group: Healthy, with no first degree relative with migraine

Exclusion criteria:

1. Pregnancy or breastfeeding,
2. Chronic pain (except for migraine for the migraine group), neurological or psychiatric syndromes or syndromes associated with pubertal maturation
3. Use of medications that impact sex hormone levels (i.e., contraceptive pills)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) response | Baseline
  This psychophysical test examine the inhibitory pain modulation efficiency. In this test, pressure pain thresholds (measures by kilopascal) are assessed before and during immersion of the foot in cold water.
Sex Hormones | Baseline
  Testosterone levels

SECONDARY OUTCOMES:
Sex hormone assessments | Baseline
  Estrogen levels
Migraine specific measures | Baseline
  Pediatric Migraine Disability Assessment (PedMIDAS) (range 0-540, higher values indicate more disability, with scores >50 considered as severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No